CLINICAL TRIAL: NCT03845725
Title: Investigation of Falls and Balance of Patients With Parkinson's Disease With Urinary Disturbance
Brief Title: Falls and Balance of Patients With Parkinson's Disease With Urinary Disturbance
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Aslıhan ÇATIKER, Principal Investigator, Ordu University
Other Study IDs: 2018-09
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Parkinson's Disease; Falls; Balance; Urinary Bladder Diseases
MeSH Terms: conditions — Parkinson Disease; Urinary Bladder Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the fall and balance conditions of Parkinson's patients according to their urinary complaints.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a slowly progressive and common neurodegenerative disease.Frequently encountered problems in lower urinary tract complaints; Bladder dysfunction, such as urinary entrapment and frequent urination.Urinary incontinence in individuals with Parkinson's disease increases the risk of falling.

The investigators will evaluate 80 patients who attended the Movement Disorders Outpatient Clinic of Ordu a University Educational Research Hospital in December 2018 and February 2019, and were diagnosed as having Parkinson's disease. Other eligibility criteria for participants were having good cognitive functions (>24 on Standardized Mini Mental Test) and were volunteers who accept to participate in the study. The investigators excluded patients that having orthopedic and / or neurological problem affecting walking and balance skills. The investigators used Unified Parkinson's Disease Rating Scale (UPDRS), modified Hoehn and Yahr Stage (H/Y), Berg Balance Scale (BBS), Falls-Efficacy Scale (FES), Timed Up and Go (TUG), and Five Times Sit to Stand Test (FTSTS), ICIQ-SF and Overactive Bladder Version-8.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease according to the United Kingdom Brain Bank diagnostic criteria
* Good cognitive functions (>24 on Standardized Mini Mental Test)
* volunteers who accept to participate in the study.

Exclusion Criteria:

* Orthopedic and / or neurological problem affecting walking or balance skills
* Not willing to participate in the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A total of 80 patients who attended the Movement Disorders Outpatient Clinic of Ordu a University Educational Research Hospital in December 2019 and February 2020 will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | Baseline
  The UPDRS is used as a gold standard reference scale. Each item is scored using a 5-point scale, where 0 means an absence of symptoms and 4 represents the worst stage
Modified Hoehn and Yahr Stage | Baseline
  The severity of PD was determined using the Modified Hoehn and Yahr Stage, which contains five stages.
  Stage 0: No signs of disease. Stage 1: Unilateral symptoms only. Stage 2: Bilateral symptoms. No impairment of balance. Stage 3: Balance impairment. Mild to moderate disease. Physically independent. Stage 4: Severe disability, but still able to walk or stand unassisted. Stage 5: Needing a wheelchair or bedridden unless assisted.
Berg Balance Scale | Baseline
  The BBS consists of 14 items and scores range from 0 (inability to perform the task) to 4 points.
Falls-Efficacy Scale | Baseline
  This scale is used to measure the perceived fear of falling. It comprises 10 questions. The score of the scale change 0-100 and the score above 70 indicates the fear of falling.
Timed Up and Go (TUG) | Baseline
  The TUG is a reliable and valid measurement tool to assess functional mobility in patients with PD
International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | Baseline
  ICIQ-SF is a short, easy-to-understand and feasible questionnaire form, which demonstrates the reliability and validity of urinary incontinence and its impact on quality of life. In ICIQ-SF questionnaire, the frequency, amount, type and effects of urinary incontinence on the daily life are questioned and scoring is performed between 0-21 values.
Overactive Bladder Version-8 | Baseline
  It is used for screening and diagnosis of overactive bladder. The BBS consists of 8 items. A total score of ≥8 indicates that the respondent may have an overactive bladder. The total score ranges from 0 to 40.

CONTACTS AND LOCATIONS:
Overall Officials: Aslıhan Çatıker, Phd, Principal Investigator — Ordu University
Locations (1):
- Movement Disorders Outpatient Clinic of Ordu a University Educational Research Hospital, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No